CLINICAL TRIAL: NCT00750178
Title: A Phase I Study Evaluating the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of MK0683 in Patients With Advanced Cancer
Brief Title: A Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of MK0683 in Patients With Advanced Cancer (0683-008)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0683-008; MK0683-008; 2008_544
Record Dates: First submitted 2008-09-08; First posted 2008-09-10 (Estimated); Last update posted 2017-04-07 (Actual); Status verified 2017-04

CONDITIONS: Cancer, Advanced
MeSH Terms: conditions — Neoplasms | interventions — Vorinostat

ARMS (1):
- A (Experimental): MK0683
  Interventions: Drug: vorinostat (MK0683 )

INTERVENTIONS:
Drug: vorinostat (MK0683 ) — Panel A: vorinostat 400 mg capsules once daily on Days 1, 5, 7-28
  Total treatment period is 28 days
  Other Names: Zolinza

SUMMARY:
This study will evaluate the safety, tolerability, pharmacokinetics, and pharmacodynamics of MK0683 in patients with advanced cancer.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years or older
* Must agree to consume high fat meal and agree to fasting conditions
* Limit alcohol consumption

Exclusion Criteria:

* Patient has a history of drug or alcohol abuse within 5 years of start of study
* Patient is known to have HIV
* Patient has participated in another investigational study within 4 weeks of start of study
* Patient cannot stop taking certain medications or herbal remedies
* Patient will require immunologic, radiation, surgery, or chemotherapy during the study
* Patient requires frequent blood transfusions
* Female patient is pregnant or nursing
* Patient has an active Hepatitis B or C infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2004-11-01 (Actual); Primary Completion 2005-08-01 (Actual); Study Completion 2005-11-01 (Actual)

PRIMARY OUTCOMES:
Safety, tolerability, and PK of MK0683 | 28 Days

SECONDARY OUTCOMES:
Urinary excretion of MK0683 | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Result] Rubin EH, Agrawal NG, Friedman EJ, Scott P, Mazina KE, Sun L, Du L, Ricker JL, Frankel SR, Gottesdiener KM, Wagner JA, Iwamoto M. A study to determine the effects of food and multiple dosing on the pharmacokinetics of vorinostat given orally to patients with advanced cancer. Clin Cancer Res. 2006 Dec 1;12(23):7039-45. doi: 10.1158/1078-0432.CCR-06-1802. PMID 17145826
- Available data/document: CSR Synopsis Links — http://www.merck.com/clinical-trials/policies-perspectives.html